CLINICAL TRIAL: NCT02208284
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study To Assess The Safety, Tolerability, And Pharmacokinetics Of Single Escalating Oral Doses Of Pf-06427878 Co-administered With Meal In Healthy Adult Subjects
Brief Title: A Single Oral Dose Study Of PF-06427878 In Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: B7871001
Record Dates: First submitted 2014-07-30; First posted 2014-08-05 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Healthy
Keywords: Single Ascending Dose; healthy subjects; Hyperlipidemia; Lipid Metabolism Disorders; Metabolic Diseases
MeSH Terms: conditions — Hyperlipidemias; Lipid Metabolism Disorders; Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1-PF-06427878 or placebo (Experimental): Single ascending doses of PF-06427878 or placebo to investigate the safety, tolerability, and PK.
  Interventions: Drug: PF-06427878; Drug: Placebo
- Cohort 2-PF-06427878 or placebo (Experimental): Single ascending doses of PF-06427878 or placebo to investigate the safety, tolerability, and PK.
  Interventions: Drug: PF-06427878; Drug: Placebo
- Cohort 3-PF-06427878 or placebo (Experimental): Single ascending doses of PF-06427878 or placebo to investigate the safety, tolerability, and PK.
  Interventions: Drug: PF-06427878; Drug: Placebo

INTERVENTIONS:
Drug: PF-06427878 — PF-06427878 or placebo will be administered once in each period as an extemporaneously prepared suspension.
  Arms: Cohort 1-PF-06427878 or placebo
Drug: Placebo — PF-06427878 or placebo will be administered once in each period as an extemporaneously prepared suspension.
  Arms: Cohort 1-PF-06427878 or placebo
Drug: PF-06427878 — PF-06427878 or placebo will be administered once in each period as an extemporaneously prepared suspension.
  Arms: Cohort 2-PF-06427878 or placebo
Drug: Placebo — PF-06427878 or placebo will be administered once in each period as an extemporaneously prepared suspension.
  Arms: Cohort 2-PF-06427878 or placebo
Drug: PF-06427878 — PF-06427878 or placebo will be administered once in each period as an extemporaneously prepared suspension.
  Arms: Cohort 3-PF-06427878 or placebo
Drug: Placebo — PF-06427878 or placebo will be administered once in each period as an extemporaneously prepared suspension.
  Arms: Cohort 3-PF-06427878 or placebo

SUMMARY:
PF-06427878 is a new compound proposed for the treatment of hyperlipidemia. The primary purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of single oral doses of PF-06427878 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non childbearing potential.
* Body Mass Index (BMI) of 17.5 to 35.4 kg/m2; and a total body weight >50 kg
* Subjects with fasting TG level of >=90 mg/dL and <=500 mg/dL following an overnight fast

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Assessment of adverse events (AEs). | 0-48 h post dose
Assessment of clinical laboratory tests. | 0-48 h post dose
Assessment of vital signs (including blood pressure and pulse rate). | 0-48 h post dose
Assessment of cardiac conduction intervals as assessed via 12-lead electrocardiogram (ECG). | 0-48 h post dose

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for PF-06427878 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours post dose
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - inf)] for PF-06427878 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours post dose
  AUC (0 - inf)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - inf). It is obtained from AUC (0 - t) plus AUC (t - inf).
Maximum Observed Plasma Concentration (Cmax) for PF-06427878 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours post dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) for PF-06427878 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours post dose
Apparent Oral Clearance (CL/F) for PF-06427878 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours post dose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) for PF-06427878 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours post dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Plasma Decay Half-Life (t1/2) for PF-06427878 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours post dose
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7871001&StudyName=A%20Single%20Oral%20Dose%20Study%20Of%20PF-06427878%20In%20Healthy%20Adult%20Subjects%20